CLINICAL TRIAL: NCT04567927
Title: Prevalence and Risk Factors for Venous Thromboembolic Events in Critically Ill Patients With SARS-CoV-2 Infection
Brief Title: Prevalence and Risk Factors for Venous Thromboembolic Events in Critically Ill Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Chiesa Alessandro Felice (Other)
Responsible Party: Sponsor-Investigator, Chiesa Alessandro Felice, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Other Study IDs: 2020-01266
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: SARS Virus
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasonography — Venous compression ultrasonography using real-time B-mode and colour doppler in transverse and longitudinal views

SUMMARY:
The purpose of the study is to assess the frequency of the occurrence of a venous thrombosis in patients with the new Coronavirus disease, who are admitted to the Intensive Care Unit for impending respiratory failure requiring intubation and mechanical ventilation. Furthermore, the investigators aim at identifying potential risk factors for thrombosis and death.

DETAILED DESCRIPTION:
Symptomatic infection with the severe acute respiratory syndrome coronavirus 2 ranges from mild to critical spectrum. About 80% of laboratory confirmed infections presented with mild symptoms, usually not requiring hospitalization. Critical disease requiring respiratory and/or circulatory support was reported in 5% of the subjects. Acute respiratory distress syndrome represents the most common complication in patients with severe disease. Several cases of venous thromboembolism in patients with laboratory confirmed infection have been reported, but it is unclear if this occurrence is higher in this specific patients' population. The purpose of the present study is to assess the prevalence of deep venous thrombosis in patients infected with SARS-CoV-2 admitted to the Intensive care Unit requiring invasive mechanical ventilation using vein ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the Intensive Care Unit
* laboratory confirmed SARS-CoV-2 infection
* invasive respiratory support

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients with laboratory confirmed SARS-CoV-2 infection admitted to the Intensive Care Unit requiring invasive respiratory support
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Period prevalence of deep vein thrombosis (DVT) | From date of inclusion in the study until the date of development of a DVT, date of death from any cause, or date of discharge from the ICU, whichever came first, assessed up to 3 months
  Percent (%) of patients with a DVT

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regionale di Bellinzona e Valli, Bellinzona, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Result] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Result] Wang T, Chen R, Liu C, Liang W, Guan W, Tang R, Tang C, Zhang N, Zhong N, Li S. Attention should be paid to venous thromboembolism prophylaxis in the management of COVID-19. Lancet Haematol. 2020 May;7(5):e362-e363. doi: 10.1016/S2352-3026(20)30109-5. Epub 2020 Apr 9. No abstract available. PMID 32278361